CLINICAL TRIAL: NCT03246191
Title: Screening and Assessing the Risk Factors and Complications of Chronic Kidney Disease：a Cross - Sectional Study
Brief Title: Screening and Assessing the Risk Factors and Complications of Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Other Study IDs: 2015BAI12B06-2
Record Dates: First submitted 2017-06-13; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, whole blood，urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample collection — blood sample collection

SUMMARY:
The study is an observational, cross-sectional study aimed at screening and accessing risk factors and complications for Chinese chronic kidney disease (CKD) patients. To investigate the prevalence of hypertension, cardiovascular and cerebrovascular diseases, protein energy malnutrition（PEM）, cognitive impairment and other complications in the CKD patients. To develop biomarkers of CKD.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* clinical diagnosis of CKD
* signed informed consent

Exclusion Criteria:

* End-stage renal disease(ESRD) or dialysis
* Acute kidney injure(AKI)
* history of solid organ or bone marrow transplantation
* active malignancy within 24 months prior to screening or metastatic cancer
* HIV infection or AIDS
* acute inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CKD complications | baseline
  hypertension, cardiovascular and cerebrovascular diseases, protein energy malnutrition(PEM), cognitive impairment
Biomarkers of kidney function | baseline

SECONDARY OUTCOMES:
Genetic analyses | baseline
  circulating microRNA
Questionnaire assessing cognitive function | baseline
  Montreal Cognitive Assessment-Basic Chinese Version
Questionnaire assessing depression | baseline
  Beck Depression Inventory scores
Questionnaire assessing risk of malnutrition | baseline
  Malnutrition-Inflammation Score
Questionnaire assessing dietary intake | baseline
  Food Frequency Questionnaire
Questionnaire assessing quality of life | baseline
  Activity of daily living（ADL）and kidney disease quality of life （KDQOLTM-36）

CONTACTS AND LOCATIONS:
Overall Officials: xiangmei chen, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No